CLINICAL TRIAL: NCT03982563
Title: Evaluating the Acceptability and Efficacy of Computerized Single-Session Interventions for Indian Adolescents
Brief Title: Computerized Single-Session Interventions for Indian Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Sangath (Other)
Responsible Party: Principal Investigator, Akash Wasil, Graduate Student, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 24922
Record Dates: First submitted 2019-06-05; First posted 2019-06-11 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Well-being; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Growth Mindset (Experimental)
  Interventions: Behavioral: Growth Mindset
- Gratitude (Experimental)
  Interventions: Behavioral: Gratitude
- Behavioral Activation (Experimental)
  Interventions: Behavioral: Behavioral Activation
- Study Skills (Sham Comparator)
  Interventions: Behavioral: Study Skills

INTERVENTIONS:
Behavioral: Growth Mindset — Reading and writing activities designed to instill the belief that people can change.
  Arms: Growth Mindset
Behavioral: Gratitude — Reading and writing activities designed to practice noticing and appreciating good things in life.
  Arms: Gratitude
Behavioral: Behavioral Activation — Reading and writing activities designed to identify and schedule positive activities.
  Arms: Behavioral Activation
Behavioral: Study Skills — Reading and writing activities designed to learn evidence-based study strategies.
  Arms: Study Skills

SUMMARY:
The overall aim of this project is to understand if single-session interventions are acceptable, culturally appropriate, and effective for Indian adolescents. The investigators will be examining the effects of three interventions on the well-being and mental health of adolescents. The investigators hypothesize that at least one of the three interventions will yield statistically significant improvements in wellbeing and mental health relative to a study skills control condition.

ELIGIBILITY:
Inclusion Criteria:

* Attending a participating secondary school
* Age 12 to 18
* Literate in English

Exclusion Criteria:

* Unable to provide informed consent

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 958 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Change in The Warwick-Edinburgh Mental Wellbeing Scale | Baseline, 4 week follow-up, 12 week follow-up
  Well-being questionnaire. Total score ranges from 14 to 70. Higher values indicate a better outcome.
Intervention Appropriateness Measure | Immediately post-intervention (i.e., 0 weeks)
  Questionnaire measuring the appropriateness of an intervention. Appropriateness refers to the perceived fit or relevance of an intervention. The total score ranges from 4 to 20. Higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | Baseline, 4 week follow-up, 12 week follow-up
  Depression Questionnaire. The total score ranges from 0 to 27. Lower scores indicate a better outcome.
Generalized Anxiety Disorder Screener-7 | Baseline, 4 week follow-up, 12 week follow-up
  Anxiety Questionnaire. The total score ranges from 0 to 21. Lower scores indicate a better outcome.
The EPOCH Measure of Adolescent Well-being | Baseline, 4 week follow-up, 12 week follow-up
  Questionnaire with five subscales measuring engagement, perseverance, optimism, connectedness, and happiness. Each subscale score ranges from 4 to 20. Higher scores indicate a better outcome. The happiness and optimism subscales will be used as secondary outcomes for this trial. A total score is not computed.
Acceptability of Intervention Measure | Immediately post-intervention (i.e., 0 weeks)
  Questionnaire measuring the acceptability of an intervention. Acceptability refers to the perception that a given treatment is agreeable or satisfactory. The total score ranges from 4 to 20. Higher scores indicate a better outcome.
Feasibility of Intervention Measure | Immediately post-intervention (i.e., 0 weeks)
  Questionnaire measuring the feasibility of an intervention. Feasibility refers to the degree to which a treatment can be successfully implemented in a given setting. The total score ranges from 4 to 20. Higher scores indicate a better outcome.
Perceived Stress Scale-4 | Baseline, 4 week follow-up, 12 week follow-up
  Questionnaire measuring perceived stress. The total score ranges from 0 to 16. Lower scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rob DeRubeis, PhD, Study Director — University of Pennsylvania; Sachin Shinde, PhD, Study Director — Sangath; Sadhana Natu, PhD, Study Director — Modern College Pune; Akash Wasil, Principal Investigator — University of Pennsylvania
Locations (4):
- India (4):
  - Dr. Kalmadi Junior High School, Pune, Maharashtra
  - The Orchid School, Pune, Maharashtra
  - JM Rathi English School, Roha, Maharashtra
  - Modern College Pune, Pune

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schleider J, Weisz J. A single-session growth mindset intervention for adolescent anxiety and depression: 9-month outcomes of a randomized trial. J Child Psychol Psychiatry. 2018 Feb;59(2):160-170. doi: 10.1111/jcpp.12811. Epub 2017 Sep 18. PMID 28921523
- [Background] Seligman ME, Steen TA, Park N, Peterson C. Positive psychology progress: empirical validation of interventions. Am Psychol. 2005 Jul-Aug;60(5):410-21. doi: 10.1037/0003-066X.60.5.410. PMID 16045394
- [Background] Emmons RA, McCullough ME. Counting blessings versus burdens: an experimental investigation of gratitude and subjective well-being in daily life. J Pers Soc Psychol. 2003 Feb;84(2):377-89. doi: 10.1037//0022-3514.84.2.377. PMID 12585811
- [Background] Chorpita BF, Becker KD, Daleiden EL. Understanding the common elements of evidence-based practice: misconceptions and clinical examples. J Am Acad Child Adolesc Psychiatry. 2007 May;46(5):647-52. doi: 10.1097/chi.0b013e318033ff71. No abstract available. PMID 17450056